CLINICAL TRIAL: NCT00390039
Title: Randomized, Double-Blind, Active- and Placebo-Controlled Study of Analgesic Efficacy and Safety of Repeated Dosing of MNS075 (Intranasal Morphine), IV Morphine, and Placebo in Acute Post-Operative Pain After Elective Orthopedic Surgery
Brief Title: Efficacy and Safety of Intranasal Morphine for Pain After Elective Orthopedic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR-003
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Pain, Postoperative
Keywords: Pain, postoperative; Surgery, orthopedic; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- A (Experimental): MNS075 7.5mg
  Interventions: Drug: Intranasal Morphine
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- C (Active Comparator): IV Morphine
  Interventions: Drug: IV morphine
- E (Experimental): MNS075 15mg
  Interventions: Drug: Intranasal morphine
- D (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- F (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Morphine — MNS075 7.5mg q1h PRN
  Arms: A
Drug: Placebo — IN Placebo q1h PRN
  Arms: B
Drug: IV morphine — IV morphine 7.5mg q3h PRN
  Arms: C
Drug: Placebo — IV Placebo q3h PRN
  Arms: D
Drug: Intranasal morphine — MNS075 15mg q3h PRN
  Arms: E
Drug: Placebo — IN Placebo q3h PRN
  Arms: F

SUMMARY:
Multiple-center, multiple-dose, randomized, double-blind, six-arm, active- and placebo-controlled study in patients with moderate to severe post-surgical pain from elective orthopedic surgery with safety observed for a total of 30 hours post first dose.

DETAILED DESCRIPTION:
Multiple-center, multiple-dose, randomized, double-blind, six-arm, active- and placebo-controlled study of repeated intermittent PRN dosing for 24 hours of Intranasal (IN) Morphine Nasal Spray (MNS075) 7.5 mg and 15 mg, 7.5 mg IV morphine infusions and placebo (either IN or IV), in patients with moderate to severe post-surgical pain from elective orthopedic surgery with safety observed for a total of 30 hours post first dose.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Scheduled (within two weeks of the screening visit) to undergo elective orthopedic surgery (e.g., bunionectomy, arthroscopic knee surgery, rotator cuff repair)
* Moderate to severe pain within 8 hours following completion of the required surgery

Exclusion Criteria:

* Previous anaphylactic or serious allergic reaction to shellfish or opioids
* History of sleep apnea

Other Inclusion/Exclusion Criteria May Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2006-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Sum of the Pain Intensity Differences (SPID) over 0-24 hours based on Visual Analog Scale (VAS) | Multiple

SECONDARY OUTCOMES:
Other measures of pain | Multiple

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmacueticals
Locations (7):
- United States (7):
  - Arizona Research Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Vertex Clinical Research, Bakersfield, California
  - University Orthopedics Center, State College, Pennsylvania
  - SCIREX Corporation, Austin, Texas
  - SCIREX Corporation, San Marcos, Texas
  - Jean Brown Research, Salt Lake City, Utah